CLINICAL TRIAL: NCT05145686
Title: The Role of Matrix Metalloproteinases on the Primary Teeth Pulpotomy Treatments With MTA and Biodentine
Brief Title: The Role of Matrix Metalloproteinases on the Primary Teeth Pulpotomy Treatments
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilsah Cogulu, Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ege U.Eth. Com.16-7/14
Record Dates: First submitted 2021-11-09; First posted 2021-12-06 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Reversible Pulpitis
Keywords: MTA; Biodentine; Pulpotomy; Matrix metalloproteinase

STUDY DESIGN:
Intervention Model Description: Experimental: Biodentine Dental materials
  Interventions:
  Drug: Biodentine Drug: ProRoot (Aggregate) Experimental: ProRoot MTA Dental Materials
  Interventions:
  Drug: Biodentine Drug: ProRoot (Aggregate)
Who Masked: Outcomes Assessor
Masking Description: observers were blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparing MMP-2, -8, -9 in reversible and irreversible pulpitis (Experimental): The coronal pulp samples from both reversible and irreversible groups were placed in an eppendorf tube containing TriPure Reagent transport medium. The MMP-2, -8 and -9 expression levels were determined with specific primers by real time polymerase chain reaction method (RT-PCR).
  Interventions: Diagnostic Test: Matris metalloproteinase -2, -8, -9 expressions
- Comparing the clinical success of MTA and Biodientine in primary molar pulpotomy treatments (Active Comparator): In reversible pulpitis group MTA (ProRoot MTA,white) was used in 21 teeth and Biodentine was used in the other 21 teeth for pulpotomy treatments. Final restorations were performed with stainless steel crowns in both group. At the end of 3, 6 and 9 months, all teeth were evaluated clinically and radiographically based on AAPD criteria: (1) absence of spontaneous pain and/or sensitivity to pressure; (2) absence of sinus, fistula, edema, and/or abnormal mobility; (3) absence of radiolucency at the interradicular and/or periapical regions; (4) absence of internal or external root resorption.
  Interventions: Diagnostic Test: Matris metalloproteinase -2, -8, -9 expressions

INTERVENTIONS:
Diagnostic Test: Matris metalloproteinase -2, -8, -9 expressions — . The aims of this in vivo study was to compare the expression levels of MMP-2, -8 and -9 in primary molars with reversible and irreversible pulpitis and to compare the clinically and radiographically success of MTA and Biodentine materials at the end of 18 months.
  Other Names: MTA and Biodentine

SUMMARY:
Matrix metalloproteinases (MMPs) are important zinc enzyme group that responsible for reducing extracellular matrix components. It has been reported that MMPs play an important role in pulpal inflammation. The aims of this in vivo study was to compare the expression levels of MMP-2, -8 and -9 in primary molars with reversible and irreversible pulpitis and to compare the clinically and radiographically success of MTA and Biodentine materials at the end of 18 months.

DETAILED DESCRIPTION:
A total of 63 mandibular primary second molar teeth of 57 healthy and cooperative children aged between 5-10 years were included in this study. The Ethical Committee of the Medical Faculty of Ege University approved the study (Reference No: 16-7/14). Detailed treatment plan was explained to the children and the parents and written informed consents were obtained.

Periapical radiographs were obtained pre-operatively. Patients with a tooth showing clinical or radiographic evidence of a deep carious lesion extending close or into the pulp chamber were considered for potential inclusion.

The teeth were assigned to different groups according to the clinical diagnosis. The diagnosis were based on strict clinical and radiographic criteria. When the dental pulp was exposed during caries removal, the following clinical and radiographic diagnostic criteria were applied; Group I (teeth with reversible pulpitis): Slight clinical symptoms of minor intensity, slightly exaggerated reaction to cold or sweet stimuli, no history of pain, no sensitivity to chewing or percussion, bleeding time from the exposed pulp tissue less than 5 minutes, and no widening of the periodontal ligament space. In pulpotomy group teeth with pulpal exposure smaller than a pinpoint, teeth with purulent/viscous, dark colored exudate detected at the exposure site, and necrotic teeth were excluded.

Group II (teeth with irreversible pulpitis): Spontanous pain, sensitivity to chewing or percussion, bleeding time from the exposed pulp tissue more than 5 minutes, and widening of the periodontal ligament space, periapical lesion.

For ethical reasons, there was no control group with blood samples from healthy caries-free teeth. All primary molars were distributed between the two treatment groups as pulpotomy (Group I, n=42) and pulpectomy (Group II, n=21).

The pulpotomy procedures and all sampling were performed by the same operator (H.E.G.) following the procedure as follows: local anesthesia (2% lidocaine (1:000,000)-Jetokain Simplex, Adeka, Turkey) was administered, and teeth were isolated by a rubberdam (Roeko Dental Dam, Coltane, Whaledent, Germany). The carious dentin was removed from the cavity, working from the periphery towards the center using a low-speed round bur (no:4). The roof of the pulp chamber was removed, and coronal pulp tissue was taken using a sharp excavator. All pulp samples were placed in 1 ml Tri Pure Reagent transport medium in pre-weighed Eppendorf tubes. The samples were weighed again and the weights were noted before storing at -80°C until the laboratory procedures. In pulpectomy group (Group II), all sampling procedures were performed as same in pulpotomy group.

In Group I, after removal of the coronal pulp, the cavity was irrigated with sterile saline, and initial bleeding was controlled by placing sterile cotton pellets moisturized with saline over the radicular pulp stump exerting slight pressure and waiting for 5 min. The teeth for which hemostasis at the canal orifices could be achieved in 5 min were included to this group. The randomization was performed as two groups in a 1 : 1 ratio by using free online software (http://www.random.org). Following the randomization procedure, patients were assigned sequential numbers in the order of enrolment and the operator was informed about the material, either with MTA (n=21) or with Biodentine (n=21).

MTA Group: According to the manufacturer's instructions, MTA (Pro Root White MTA, Dentsply, Tulsa Dental Specialties, USA) powder was mixed with sterile water in a 3:1 powder/water ratio to obtain a thick creamy paste, then placed on the floor of the pulp chamber. The MTA mixture was covered with a moistened cotton pellet and then temporarily sealed using glass ionomer cement (GIC-Ketac Molar Easymix, 3M Espe, Seefeld, Germany) until the second visit.

Biodentine Group: Biodentine (Septodont, Saint-Maur-des-Fossés, France) capsule was gently tapped on a hard surface to diffuse powder, five drops of liquid from the single dose dispenser were poured into the capsule and then mixed with 4200 rpm 30 seconds and placed over the pulp stumps using an appropriate spatula advised by the manufacturer. After allowing Biodentine to set for 12 min, the teeth were temporarily sealed with GIC as same in MTA group.

After 24 hours, the teeth in both groups were restored with preformed stainless -steel crowns (3M Espe, Stainless Steel Crowns, Seefeld, Germany). The participants were recalled at 6, 12 and 18 months after the treatment. At each follow-up visit, clinical and radiographic examinations were performed by two calibrated blinded examiners. All teeth were evaluated clinically and radiographically according to the criteria: (1) absence of spontaneous pain and/or sensitivity to pressure, (2) absence of sinus, fistula, edema, and/or abnormal mobility, (3) absence of radiolucency at the interradicular and/or periapical regions, (4) absence of internal or external root resorption. The absence of spontaneous pain, pathologic mobility, tenderness to percussion, swelling, fistula, and gingival inflammation was considered as a clinical success, whereas the absence of internal/external root resorption and periapical/furcal radiolucency was considered as a radiographic success. Calcific metamorphosis of the pulp was not considered as a failure.

Pulp tissue was washed in phosphate-buffered saline (Gibco, Invitrogen, Karlsruhe, Germany) for 1 min, cut into small pieces, transferred to cell-culture plates and incubated with Dulbecco's modified Eagle's medium containing 10% fetal bovine serum (Gibco BRL, Life Technologies, Grand Island, NY, USA), penicillin-G (100 U⋅mL), streptomycin (100 µg⋅mL) and Fungizone (0.25 g⋅mL) (GeminiBio-Products Inc., Woodland, CA, USA) at 37 °C in a humidified atmosphere of 5% CO2. Migration of cells from the pulpal tissue occurred 1 week later, and cultures were established and maintained in standard culture medium. Medium was refreshed three times per week, and cells were split, after reaching confluence. Pulp cells between the third and eighth passages were used in this study (ref).

RNA was extracted from the treated cells using RNAiso Plus (TaKaRa Bio, Shiga, Japan). cDNA was synthesized from 400 ng of total RNA using the PrimeScript RT reagent kit (TaKaRa Bio, Otsu, Japan) according to the manufacturer's instructions. One-tenth of the cDNA obtained was added for a final volume of 20 µL for each reaction containing SYBR Green I (TaKaRa Bio, Shiga, Japan). The primers for MMP-2, -8 and -9 were as follows (sense/antisense):

MMP-2: 5'-ATC CTG GCT TTC CCA AGC TC-3'/3'-CAC CCT TGA AGA AGT AGC TGT G-5'. MMP-8:5'-CTGTTGAAGGCCTAGAGCTGCTGCTCC3'/5'CATCTTCTCTTCAAACTCTACCC-3'. MMP-9: 5'-GGG CTT AGA TCA TTC CTC AGT G-3'/3'-GCC ATT CAC GTC GTC CTT AT-5'. (ref) Reactions were run on an ABI Step One real-time PCR system (Applied Biosystems, Foster City, CA, USA) with the following program: 45 cycles of 95 °C for 10 s, 60 °C for 15 s and 72 °C for 20 s. For relative comparisons of each gene, the investigators analysed the threshold cycle (Ct) value of the real-time PCR data using the 2-ΔΔCt method.20 The PCR products were analyzed on a 1.5% agarose gel containing 1 pg/mL ethidium bromide, which attaches to nucleic acids, allowing the PCR products to be visualized under UV light. The gel was photographed to allow the products to be quantitated as described below. After finding the linear portion for each set of primers for quantitation of the products, the investigators quantitated the products with an image processing and analyzing program (ScionImage PC, Scion Corporation, Frederick, MD, USA) to analyze the expression of MMP-2, -8 and -9.(ref) Statistical Analysis The statistical analysis was performed using SPSS for Windows version 25.0 (SPSS, Chicago, IL, USA). A p-value of <0.05 was considered to be statistically significant.

Data were analysed using a Fisher Exact Test in addition to chi-square tests to perform inter- and intra- group comparisons, respectively.

The Fisher's Exact Test was used for testing the levels of MMP-2, -8, -9 expression between the reversible and irreversible pulpitis groups.

The 6, 12 and 18 months clinically and radiographically success of MTA and Biodentine materials were tested by chi-square test.

Mann Whitney U test was used in comparing the MMP-2, -8, -9 expressions between successful and failed pulpotomy groups.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative pediatric patients aged 5-10 years,
* Deep carious lesion in mandibular primary second molars,
* The subjects did not receive any antiinflammatory medication 3 months prior to the study,
* Feasible restorative treatment,
* Positive parental informed consent.

Exclusion Criteria:

* Uncooperative children,
* Children with medically compromised disease,
* Presence of pathological root resorption and/or bone defect,
* Physiological root resorption more than one-third of the root,
* Unrestorable teeth,
* Negative parental informed consent.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — 50% boy, 50% girl
Enrollment: 57 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The role of MMP-2, 8 and 9 in reversible and irreversible pulpitis | 18 months
  The expression levels of MMP-2, 8 and 9 were detected
Comparison of the clinical and radiographic success of MTA and Biodentine in primary teeth pulpotomy treatment | 18 months
  MTA and Biodentine materials were used in primary molars with reversible pulpitis. At the end of 6, 12 and 18 months, all teeth were evaluated clinically and radiographically based on AAPD criteria: (1) absence of spontaneous pain and/or sensitivity to pressure; (2) absence of sinus, fistula, edema, and/or abnormal mobility; (3) absence of radiolucency at the interradicular and/or periapical regions; (4) absence of internal or external root resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Dilşah Çoğulu, Prof. Dr., Principal Investigator — Ege University, Izmir, Turkey
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Gerihan HE, Cogulu D, Oncag O, Durmaz A, Kuru EH. Assessment of MMP levels in reversible and irreversible pulpitis and a randomized controlled trial comparing clinical success of two different calcium-silicate cements in pulpotomy treatment of primary molars with an 18-month follow-up. BMC Oral Health. 2024 Aug 30;24(1):1020. doi: 10.1186/s12903-024-04795-5. PMID 39215293